CLINICAL TRIAL: NCT02517853
Title: Prospective and Randomized Study to Evaluate the Efficiency of Percutaneous Neurostimulation of Posterior Tibial Nerve in the Treatment of Low Anterior Resection Syndrome (LARS)
Brief Title: Efficiency of Neurostimulation of Tibial Nerve in the Treatment of Low Anterior Resection Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NETP-01-2014
Record Dates: First submitted 2015-07-28; First posted 2015-08-07 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Colorectal Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tibial nerve stimulation (Experimental): Tibial nerve stimulation during 16 sessions
  Interventions: Device: Posterior tibial nerve stimulation
- Sham comparator (Sham Comparator): Sham tibial nerve stimulation during 16 sessions
  Interventions: Device: Sham posterior tibial nerve stimulation

INTERVENTIONS:
Device: Posterior tibial nerve stimulation
  Arms: Tibial nerve stimulation
Device: Sham posterior tibial nerve stimulation
  Arms: Sham comparator

SUMMARY:
The aim of this study is to evaluate the efficiency of the Neuroestimulation of the Posterior Tibial Nerve for the treatment of this syndrome.

A multicentric, prospective, randomized study will be performed in patients affected with severe LARS symptoms. Patients will be randomized in two groups:

1. Control group- placebo
2. Treatment group: neuroestimulation of the posterior tibial nerve

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and under 75 years who have been undergone anterior resection of the rectum with sphincter preservation for rectal cancer
* Patients with LARS score > 29

Exclusion Criteria:

* Patient with intestinal inflammatory disease
* Patients with known irritable colon disease
* Pregnancy patients
* Patients with others intestinal resection segments different from the rectum
* Patients with metastatic disease
* Patient with previous history of posterior tibial neurostimulation or sacral nerve stimulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2019-08-07 (Actual)

PRIMARY OUTCOMES:
Tibial nerve stimulation efficacy measured by LARS score | 1 month
Tibial nerve stimulation efficacy measured by LARS score | 3 months
Tibial nerve stimulation efficacy measured by LARS score | 6 months
Tibial nerve stimulation efficacy measured by LARS score | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Vall d'Hebron, Barcelona

REFERENCES:
- [Derived] Marinello F, Planellas P, Fraccalvieri D, Ortega-Torrecilla N, Gil J, Kreisler E, Pellino G, Espin-Basany E. Exploratory Analysis of Urinary and Sexual Dysfunction in Patients With Low Anterior Resection Syndrome Undergoing Sacral Neuromodulation: Insights From the SANLARS Trial. Dis Colon Rectum. 2026 Feb 1;69(2):226-234. doi: 10.1097/DCR.0000000000004050. Epub 2025 Nov 18. PMID 41538382
- [Derived] Marinello F, Fraccalvieri D, Planellas P, Adell Trape M, Gil JM, Kreisler E, Pellino G, Espin-Basany E. Sacral Neuromodulation in Patients With Low Anterior Resection Syndrome: The SANLARS Randomized Clinical Trial. Dis Colon Rectum. 2024 Mar 1;67(3):435-447. doi: 10.1097/DCR.0000000000003143. Epub 2023 Dec 11. PMID 38084933
- [Derived] Marinello FG, Jimenez LM, Talavera E, Fraccalvieri D, Alberti P, Ostiz F, Frago R, Blanco A, Pellino G, Espin-Basany E. Percutaneous tibial nerve stimulation in patients with severe low anterior resection syndrome: randomized clinical trial. Br J Surg. 2021 Apr 30;108(4):380-387. doi: 10.1093/bjs/znaa171. PMID 33793754